CLINICAL TRIAL: NCT06632678
Title: PPI in the Design and Conduct of Non-pharmacological, Non-commercial Spanish Clinical Trials Completed and Published in 2009-2024
Brief Title: Patient and Public Involvement (PPI) in Non-pharmacological, Non-commercial Spanish Clinical Trials
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Rafael Dal-Ré, Emeritus investigator, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Other Study IDs: IIS-FJD-RDR-2024-001
Record Dates: First submitted 2024-10-01; First posted 2024-10-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-12

CONDITIONS: Any Condition
MeSH Terms: interventions — Diet; Exercise; Educational Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

INTERVENTIONS:
Other: behavior, procedure, diet, exercise, device, education, and any other — Any type of intervention except pharmacological interventions (drugs, biologicals, genetics)

SUMMARY:
Patient and public involvement (PPI) in the design and conduct of clinical trials has been encouraged for many years. Yet, there is no data available describing how many trials sponsored by non-commercial Spanish individuals or organizations have liaised with patients, relatives or caregivers and the public to consider their preferences and values in the design of trials assessing non-pharmacological interventions.

DETAILED DESCRIPTION:
This systematic review will be conducted in clinical trial registers that host non-pharmacological trials.

PPI is not an item of the information included on clinical trial registers. Thus, the objective of this study is to describe the percentage of non-pharmacological non-commercial Spanish trials with PPI as reported in published reports. For this reason our interest is on trials that have been completed. The published reports of interest are those that first described main trial results; those describing trial protocols. In the abscence of peer-reviewed reports, preprints will be considered. No other type of reports will be considered as valid source of information.

The study will review the trials (i.e.,interventional studies) conducted in Spain, and completed between September 01, 2009 and September 01, 2024. Five registers will be reviewed: clinicaltrials.gov, ISRCTN, DRKS, REBEC, and ACTRN. It is assumed that most of non-pharmacological non-commercial Spanish-sponsored trials will be registered in these five registers as per the information gathered from a previous study on COVID-19 Spanish non-commercial trials. The published reports of all completed trials from these four registers will be searched on PubMed and Google Scholar by using the trials IDs. Corresponding authors will be contacted only in the case it is impossible to retrieve the article or preprint.

In addition to PPI, and to characterize the trials, several variables will be also captured from the articles such as trial design, number of participants, condition/indication, type of intervention, year of publication, number of citations, citations/year, whether the trial was conducted following the Declaration of Helsinki proisions, whether all authors were non-physicians, and data availability statement. In addition, where was the trial registered. We will also register the Spanish region where the sponsor was located, information that will only be used in case it is deem necessary. In other words, the information to be gathered should be captured from the published reports.

ELIGIBILITY:
Inclusion Criteria: Spanish sponsor; non-commercial sponsor. -

Exclusion Criteria: trials assessing pharmacologic interventions.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy and patients with any disease or condition
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Patient and public involvement | Published report; Day 1
  Presence of a PPI statement in the published report

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Dal-Ré, MD, PhD, MPH, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Locations (2):
- Spain (2):
  - University Hospital Fundación Jimenez Diaz, Madrid
  - Hospital La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Dal-Ré R, García-Méndez E. Patient and public involvement in registered non-pharmacological non-commercial Spanish trials completed in 2009-2024: A systematic review. Medicina Clinica (Barc) 2025, 165:106964 — https://www.elsevier.es/es-revista-medicina-clinica-2-articulo-patient-public-involvement-in-registered-S0025775325001903